CLINICAL TRIAL: NCT00874263
Title: The Role of Endoscopic Confocal Microscopy in Diagnosing Colorectal Cancer and Other Gastrointestinal Pathologies in Vivo
Brief Title: Confocal Probe-based Endoscopic Imaging, Colorectal Cancer, Gastrointestinal (GI) Pathologies
Acronym: ASGE-FNDT-1
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other)
Responsible Party: Principal Investigator, Michael Wallace, Principal Investigator, Mayo Clinic
Other Study IDs: 07-007521; ASGE Grant#FNDT-1
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Colonic Polyps; Esophageal Diseases
Keywords: Probe-based imaging of GI pre-malignant or malignant lesions
MeSH Terms: conditions — Colonic Polyps; Esophageal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The recently developed endoscopic Confocal probe microscopy system allows imaging of surface epithelium during ongoing endoscopy (upper and lower) with the potential of immediate diagnosis of various GI pre-malignant and malignant lesions. The purpose of this study is to determine if using this new Confocal probe system can find pre-cancerous abnormalities in the stomach and colon.

Hypothesis: The confocal endomicroscopy images of colorectal lesions during the standard colonoscopies could help the classification in vivo of colorectal neoplastic and non-neoplastic lesions. This could direct further endoscopic interventions such as targeted biopsies of early colorectal cancer lesions and the endoscopic resection of such lesions during screening colonoscopies.

Primary Aim

1. To determine the key confocal image features of neoplastic and pre-neoplastic colorectal lesions including flat and raised adenomatous polyps, intraepithelial neoplasia and cancer as well as benign lesions such as hyperplastic polyps and normal colonic epithelium and to estimate which morphologic features best distinguish neoplastic and non-neoplastic tissues.

   Secondary Aims:
2. To determine the initial sensitivity and specificity of confocal microendoscopy imaging for classification of adenomatous from hyperplastic polyps of the colon.
3. In this exploratory phase of the study to develop a library of confocal microendoscopic imaging characteristics of other GI pathologies such as:

   1. Barrett's esophagus in comparison to Barrett's esophagus with dysplasia, and normal squamous esophagus.
   2. Other encountered inflammatory and neoplastic conditions within the GI tract in which biopsy or removal of tissue would routinely be indicated.

The second phase of the study will focus on establishing the sensitivities, specificities, accuracy of confocal images of colorectal lesions and other GI pathologies as well as inter-observer agreement and learning curve in interpretation of confocal images.

DETAILED DESCRIPTION:
Colorectal cancer is the second most common cause of cancer-related death in the U.S. Although removal of pre-malignant polyps has been shown to reduce the risk of colorectal cancer, up to 50% of removed colonic polyps are hyperplastic with no malignant potential. Removal of these benign polyps exposes the patient to polypectomy-related complications and cost without any benefit. Current standard endoscopes with the use of accessory confocal endomicroscopy probe will allow both routine and confocal microscopy imaging. Colonoscopies or upper endoscopies will be performed as routine including conscious sedation. A special fiber through the scope, combined with a small amount of dye called fluorescein given by vein, will be used to obtain microscopic views during the endoscopic procedure. If a colorectal lesion or other GI lesion is found that would normally require biopsy, the site of biopsy will be evaluated by confocal imaging with the Cellvizio-GI Fiberoptic probes prior to biopsy or removal of the suspicious tissue. Following image acquisition, the lesion will be biopsied or removed as per standard clinical care. Standard endoscopic variables for each lesion will be recorded including: name and record number, date, time, an exact time of fluorescein injection and time of image acquisition, lesion location, size, and suspected findings (inflammation, dysplasia, type of polyp) and final histological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 100
2. Any patient undergoing screening and/or surveillance colonoscopy and/or upper endoscopy with possible biopsy or removal of tissue by polypectomy

Exclusion Criteria:

1. Unwilling to consent
2. Allergy to fluorescein
3. Lack of any pathological state that would require biopsy at the time of endoscopy (will be considered "screen failure" since this will not be known until after consent is obtained and sedated endoscopy performed)
4. Women of child-bearing age who are sexually active and not practicing an acceptable form of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting to Mayo Clinic, Jacksonville, Florida for a screening, surveillance colonoscopy, and/or a diagnostic and surveillance upper endoscopy, will be eligible based on inclusion and exclusion criteria. Eligible patients will be offered entry into the study on the day of the procedure in the hospital GI or Mayo Clinic Jacksonville endoscopy suites.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Endoscopic Confocal microscopy may help distinguish small adenomatous polyps with malignant potential from non-neoplastic (hyperplastic) polyps in real- time enabling immediate diagnosis and removal of only polyps with truly malignant potential. | one year

SECONDARY OUTCOMES:
Endoscopic Confocal microscopy has the potential to fundamentally change the way endoscopy and pathology interact by allowing near histological-quality imaging in vivo, without the need, risk, and cost of tissue removal. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Wallace, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Andre B, Vercauteren T, Buchner AM, Krishna M, Ayache N, Wallace MB. Software for automated classification of probe-based confocal laser endomicroscopy videos of colorectal polyps. World J Gastroenterol. 2012 Oct 21;18(39):5560-9. doi: 10.3748/wjg.v18.i39.5560. PMID 23112548
- [Derived] Shahid MW, Buchner A, Gomez V, Krishna M, Woodward TA, Raimondo M, Wallace MB. Diagnostic accuracy of probe-based confocal laser endomicroscopy and narrow band imaging in detection of dysplasia in duodenal polyps. J Clin Gastroenterol. 2012 May-Jun;46(5):382-9. doi: 10.1097/MCG.0b013e318247f375. PMID 22499072
- [Derived] Buchner AM, Shahid MW, Heckman MG, Krishna M, Ghabril M, Hasan M, Crook JE, Gomez V, Raimondo M, Woodward T, Wolfsen HC, Wallace MB. Comparison of probe-based confocal laser endomicroscopy with virtual chromoendoscopy for classification of colon polyps. Gastroenterology. 2010 Mar;138(3):834-42. doi: 10.1053/j.gastro.2009.10.053. Epub 2009 Nov 10. PMID 19909747